CLINICAL TRIAL: NCT01804543
Title: Impact of Ranolazine on Myocardial Ischemia Detected by High-Field 3T Cardiovascular Magnetic Resonance (CMR) Imaging and P-31 Spectroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Westside Medical Associates of Los Angeles (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, David Gallegos, RN, Principal Investigator, Westside Medical Associates of Los Angeles
Other Study IDs: IN-US- 259-0140
Record Dates: First submitted 2012-08-03; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Angina; Heart Disease
MeSH Terms: conditions — Angina Pectoris; Heart Diseases | interventions — Ranolazine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Angina, Heart Disease: ranolazine 500 mg twice daily for 1 week, then 1000 mg twice daily for 3 weeks
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — ranolazine 500 mg, then 1000 mg twice a day
  Other Names: Ranexa

SUMMARY:
Evaluation of use of ranolazine in patients with stable heart pain with cardiac magnetic resonance imaging (CMRI) and phosphorous-31 magnetic resonance spectroscopy (31P MRS). Subsequent testing using these modalities will show improved oxygen to the heart muscle.

DETAILED DESCRIPTION:
Specific Aim:

To determine in patients with stable coronary artery disease with documented inducible ischemia, if treatment with ranolazine leads to reduced intracellular ischemia as detected by CMR perfusion imaging and 31P spectroscopy at 3 Tesla.

Abstract:

Despite many advances in cardiovascular medicine for patients with coronary artery disease (CAD), many patients in the United States continue to have the morbidity and mortality associated with chronic stable angina. Ranolazine is a novel late sodium current inhibitor shown to be effective in treating angina in patients with chronic stable coronary artery disease without affecting the blood pressure heart rate product. It has been shown to reduce myocardial energy utilization by enhancing diastolic myocardial relaxation and possibly by increasing myocardial blood flow. While ranolazine has been demonstrated to improve size and severity of stress-induced myocardial perfusion defects, it's direct effect on myocardial metabolism and cellular ischemia has not been tested in humans. We propose using cardiac magnetic resonance imaging (CMRI) and phosphorous-31 magnetic resonance spectroscopy (31P MRS) to evaluate patients with chronic stable angina before and after 4 weeks of a stable dose of ranolazine to detect changes in myocardial blood flow, ventricular function, myocardial scar and metabolic parameters of cellular ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age with stable angina pectoris or an anginal equivalent symptom (e.g. atypical chest discomfort, dyspnea, easy fatigue) AND
2. Mild, moderate or severe myocardial ischemia detected on nuclear perfusion imaging (exercise or pharmacologic SPECT or Rubidium PET), exercise stress echocardiography or stress cardiac MRI OR Documentation of obstructive coronary artery with at least one major coronary artery (left anterior descending, circumflex or right coronary artery) of at least 70% by either conventional or CT coronary angiography.

Exclusion Criteria:

1. Acute coronary syndrome including unstable angina or non ST elevation myocardial infarction within the last 60 days
2. ST-elevation myocardial infarction within 60 days
3. Equivocal myocardial ischemia on non-invasive testing or studies demonstrating reversible perfusion defects complicated by significant attenuation artifacts.
4. Recent PCI within the last 60 days
5. Recent CABG within the last 60 days
6. Inability to sign informed consent
7. Patients who have taken ranolazine within 30 days of screening
8. Patients taking strong CYP3A inhibitors e.g. ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir
9. Patients taking inducers of CYP3A e.g. rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort
10. Patients with liver cirrhosis or liver disease that is Grade B or C by the Child-Pugh Classification
11. Prior allergic reaction or intolerance to ranolazine
12. Patients with a history of inherited or acquired prolonged QT interval
13. Moderate to severe claustrophobia or previous inability to undergo an MRI exam
14. Patients with implanted pacemaker or internal cardiac defibrillator
15. Patients who have a metallic foreign body implants (metal silver in their eye, cochlear implants) or have an aneurysm clip in their brain
16. GFR < 30 ml/m2
17. Type 2 second degree heart block (Mobitz II) in the absence of functioning permanent pacemaker.
18. Sinus node dysfunction in the absence of functioning permanent pacemaker.
19. Patients taking dipyridamole therapy.
20. Active bronchospasm (active asthma or COPD with active wheezing.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with chest pain or equivalence (atypical chest pain, shortness of breath, or fatigue)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
parameters of cellular ischemia by 31P MRS | post 4 weeks of therapy with ranolazine

SECONDARY OUTCOMES:
myocardial perfusion indices | post 4 weeks of therapy with ranolazine

CONTACTS AND LOCATIONS:
Locations (1):
- Westside Medical Associates of Los Angeles, Beverly Hills, California, United States